CLINICAL TRIAL: NCT06131242
Title: The Application Value of Serum S100β in Acute Mild Traumatic Brain Injury.
Brief Title: The s100β Levels in Patients With Mild Brain Injury.
Status: Not yet recruiting | Type: Observational
Sponsor: Sumei Lu (Other)
Responsible Party: Sponsor-Investigator, Sumei Lu, Principal Investigator, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(109)
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- According to age, the group was divided into 18-45, 45-65, and > 65 years old.
  Interventions: Other: It is an observational study

INTERVENTIONS:
Other: It is an observational study — It is an observational study

SUMMARY:
Mild traumatic brain injury (TBI) accounts for the majority of TBI. At present, whether TBI has traumatic intracranial lession is mainly diagnosed by computed tomography (CT), while only 5% of mild TBI has positive CT results. The risk stratification method for patients with mild TBI is needed to reduce unnecessary CT use and reduce medical costs.

S100β is a protein in glial cells and can be used as a biomarker of brain injury. S100β is showed to have the clinical and economic value in ruling out traumatic intracranial lesions in mild TBI patients in Europe and the United States. However, it was showed to have difference between races, and there lacks systematic research data from Chinese population. In addition, if it is used for emergency departments, it is necessary to evaluate new rapid detection methods.

This study is based on a novel fast S100β test. The reference intervals of S100β in Chinese adults will be established. Further, evaluation of S100β in diagnosis of traumatic intracranial lesions in acute mild TBI will be conducted from the perspective of clinical and economic value in China, which will provide data for screening of low-risk TBI patients and avoiding unnecessary CT use in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Study on healthy people: Apparently healthy people >18 years old who came to our hospital for physical examination.
2. Study of emergency trauma patients: 1) Emergency trauma patients at least 18 years old with suspected brain injury; 2) Glasgow Coma Score 13-15 (patients with mild traumatic brain injury); 3) Closed head trauma; 4) Clinical judgment of patients requiring craniocerebral CT examination.

Exclusion Criteria:

1. Healthy population study: stroke history, trauma, surgery, mental illness, senile dementia, cognitive impairment, and tumor patients within 3 months.
2. Study of emergency trauma patients: 1) neurological or psychiatric history, 2) intellectual disabilities, 3) alcohol or drug addiction (trauma after drinking was eligible for inclusion, but alcohol consumption was recorded), 4) brain tumor patients, 5) time of trauma was not available, and 6) patients whose clinical conditions were deemed unsuitable for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy people or patients with mild traumatic brain injury.
Sampling Method: Probability Sample
Enrollment: 494 (Estimated)
Dates: Start 2023-11-09 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The serum s100β levels | 2024.6-2026.6

CONTACTS AND LOCATIONS:
Overall Officials: Sumei Lu, Study Director

IPD SHARING:
Plan to Share IPD: No